CLINICAL TRIAL: NCT00372073
Title: A Phase IIb Randomized Study of Oral Seliciclib in Patients With Previously Treated Non-Small Cell Lung Cancer
Brief Title: Efficacy Study of Oral Seliciclib to Treat Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CYC202-06-14 (A1)
Record Dates: First submitted 2006-09-03; First posted 2006-09-06 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Roscovitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 with seliciclib (Active Comparator): Oral seliciclib at 1200mg b.i.d. for 3 consecutive days as an outpatient beginning on day 1 every 2 weeks for 3 cycles as run-in. Patients (randomized) continue on treatment if derived clinical benefit during run-in period.
  Interventions: Drug: seliciclib
- Arm 2 with placebo control (Placebo Comparator): Randomized to placebo after run-in period.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: seliciclib — 1200 mg bid x 3 days every 2 weeks
  Other Names: CYC202
  Arms: Arm 1 with seliciclib
Drug: placebo — 1200 mg bid x 3 days every 2 weeks
  Arms: Arm 2 with placebo control

SUMMARY:
A phase 2 study to evaluate efficacy of oral seliciclib in treating non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
A randomized Phase II study of an experimental anti-cancer drug called seliciclib with objectives of evaluating safety and efficacy in patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with histologically-confirmed recurrent non-small cell lung cancer have had at least two prior systemic treatment regimens
* Must have measurable disease according to RECIST
* Eastern Cooperative Oncology Group performance status 0-1
* Adequate bone marrow, hepatic and renal function
* Ability to swallow capsules
* At least 3 weeks from prior systemic treatments including investigational anti-cancer therapy, at least 7 days from prior radiation therapy and have recovered from prior toxicities
* At least 3 weeks from major surgery

Exclusion Criteria:

* Non-small cell cancer histology contains a component of small cell lung cancer
* Previously untreated CNS metastasis or progressive CNS metastasis
* Prior treatment with a CDK inhibitor
* Currently receiving radiotherapy, biological therapy, or any other investigational therapy
* Uncontrolled intercurrent illness
* Having other cancers that have been treated with chemotherapy or biological therapy in the past 5 years with the exception of adequately treated in situ cervical cancer or basal cell skin cancer
* Pregnant or lactating women
* Known to be HIV-positive
* Active hepatitis B and/or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2006-08-09 (Actual); Primary Completion 2009-03-03 (Actual); Study Completion 2009-04-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | over the course of the study
  Time until the disease starts progressing

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Belani, M.D., Study Chair — Milton S. Hershey Medical Center
Locations (20):
- United States (20):
  - Arizona Cancer Center, Tucson, Arizona
  - Pacific Coast Hematology Oncology Group, Fountain Valley, California
  - Pasco Hernando Oncology, New Port Richey, Florida
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - University of Maryland, Greenebaun Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Columbia Presbyterian Medical Center, New York, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburg Cancer Institute, Pittsburgh, Pennsylvania
  - The Family Cancer Center, Collierville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
  - Center for Oncology Research and Treatment, Dallas, Texas
  - East Texas Medical Center, Tyler, Texas
  - Danville Hematology Oncology, Danville, Virginia

REFERENCES:
- [Derived] Malumbres M, Barbacid M. Cell cycle, CDKs and cancer: a changing paradigm. Nat Rev Cancer. 2009 Mar;9(3):153-66. doi: 10.1038/nrc2602. PMID 19238148